CLINICAL TRIAL: NCT07048665
Title: Effectiveness of Trans-Arterial Chemo Embolization for Hepatocellular Carcinoma on Follow-Up CT Triphasic Liver
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/906
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT Images
  Interventions: Diagnostic Test: CT Imagesa in HCCT

INTERVENTIONS:
Diagnostic Test: CT Imagesa in HCCT — Cross-sectional imaging with computed tomography (CT) scanning and magnetic resonance imaging (MRI) is most commonly used to detect hepatocellular carcinoma (HCC). CT scanning is frequently the first examination; however, MRI has superior contrast resolution and may better detect lesions less than 1 cm in diameter

SUMMARY:
"HCC is a major challenge due to greater recurrence rates and variable treatment responses. TACE is widely used, but its success relies on accurate follow-up imaging. CT Triphasic Liver Imaging plays a vital role in assessing treatment response, guiding clinical decisions, and improving patient outcomes. The purpose of this study is to investigate the relationship between response of treatment, gender, age, and the cause of HCC. The purpose of the study is to evaluate how well TACE (trans-arterial chemoembolization) works for patients with HCC.

DETAILED DESCRIPTION:
This will be a retrospective observational study aimed at evaluating the effectiveness of Trans-Arterial Chemo-Embolization in the management of Hepatocellular Carcinoma (HCC) using follow-up CT Triphasic Liver imaging. Patient records and imaging data from past cases will be reviewed to assess post- treatment tumor response and progression.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female.
* Patients diagnosed with HCC who underwent TACE.
* Patients with no portal vein tumor thrombus (PVTT) or no extra Extrahepatic Metastases at the time of initial TACE treatment.
* Patients who underwent TACE within last your years from the study start date.

Exclusion Criteria:

* Patients with incomplete or missing medical records and imaging studies.
* Patients with a history of severe comorbidities that might interfere with treatment response evaluation
* Patients who were contraindicated for CT scans at the time of follow-up.
* Patients that are contradicted with CT scan.
* Patient who underwent TACE more than four years before the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: his will be a retrospective observational study aimed at evaluating the effectiveness of Trans-Arterial Chemo-Embolization in the management of Hepatocellular Carcinoma (HCC) using follow-up CT Triphasic Liver imaging. Patient records and imaging data from past cases will be reviewed to assess post- treatment tumor response and progression.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
self admisistered questioner | 12 Months
  self-administered questionnaire for the evaluation of HCCT, having a score range from 0 to 50.
  The more the score shows that issues worsen.

CONTACTS AND LOCATIONS:
Locations (1):
- AYK Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No